CLINICAL TRIAL: NCT00417378
Title: Left Ventricular Assist Device (Impella LP 2.5) vs. Intraaortic Balloon Counterpulsation (IABP) in Patients With Cardiogenic Shock and Acute Coronary Syndromes
Brief Title: Efficacy Study of LV Assist Device to Treat Patients With Cardiogenic Shock (ISAR-SHOCK)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Abiomed Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Impella M22
Record Dates: First submitted 2006-12-29; First posted 2007-01-01 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Shock, Cardiogenic; Myocardial Infarction
Keywords: ACS
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Intraaortic balloon counterpulsation (IABP)
  Interventions: Device: Intraaortic Balloon Pump
- 2 (Experimental): Left Ventricular Assist Device (Impella LP2.5)
  Interventions: Device: Left Ventricular Assist Device Impella LP 2.5

INTERVENTIONS:
Device: Left Ventricular Assist Device Impella LP 2.5 — Left Ventricular Assist Device
  Arms: 2
Device: Intraaortic Balloon Pump — Counterpulsation
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a left ventricular assist device in comparison to a standard treatment with an intraaortic balloon pump (IABP) in patients with cardiogenic shock due to left ventricular failure following an acute coronary syndrome (myocardial infarction).

DETAILED DESCRIPTION:
Cardiogenic shock due to a left ventricular failure after myocardial infarction (MI) is associated with a mortality rate of 50-70 % despite all efforts such as immediate PCI of the occluded vessel, positive inotropic drugs, and the use of intraaortic balloon counterpulsation (IABP). While urgent heart transplantation or the surgical implantation of high-volume left ventricular assist devices are possible treatment options, a widespread use of these techniques for this common complication of myocardial infarction is limited. Because of the easy, percutaneous use of an intraaortic balloon pump, IABP is the method of choice for mechanical assistance in these patients. Despite a lack of randomized data, the ACC/AHA guidelines recommend the use of an intraaortic balloon counterpulsation (Level of evidence IB) in patients with a cardiogenic shock after myocardial infarction. However, improvement of the hemodynamic state by the use of an IABP is limited and the lack of an active cardiac support remains the major limitation of this treatment. Percutaneous left ventricular assist devices may both overcome the limitation of a surgical approach and offer the potential benefit of an active cardiac support during recovery of the failing left ventricle after PCI.

Previous studies have demonstrated a significant improvement of hemodynamic parameters by the use of a catheter-based miniaturized rotary blood pump (Impella LP2.5, Abiomed-Impella CardioSystems GmbH, Aachen, Germany), that is placed retrogradely through the aortic valve. The microaxial pump aspirates blood from the left ventricle and expels it to the ascending aorta with a maximal flow of 2.5 L/min. Randomized data comparing the LVAD with IABP are missing. Therefore, this trial will primarily compare the hemodynamic improvement of the LVAD (Impella LP2.5) with the hemodynamic improvement of an intraaortic balloon counterpulsation (IABP), while secondarily feasibility, safety and mortality will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome (ACS/AMI) < 48h and cardiogenic shock defined as:

  * Clinical criteria: Hypotension (syst.BP < 90 mmHg and HR > 90/min or an AV- Block II-III) or the need for positive inotropic drugs to maintain BB > 90mm Hg)and end-organ hypoperfusion
  * Hemodynamic criteria: CI < 2.2 L/min/qm and a PCWP > 15 mmHg or an EF of LV < 30% and LVEDP > 20 mmHg.
* Written informed consent of the patient or his/hers relatives

Exclusion Criteria:

* Age < 18 years
* Prolonged Resuscitation (> 30min)
* Hypertrophic Obstructive Cardiomyopathy
* Thrombus in left ventricle
* Treatment with IABP
* Severe valvular disease or mechanical heart valve
* Cardiogenic Shock due to mechanical complications of myocardial infarction such as VSD, acute mitral regurgitation >II°, rupture of the ventricle
* Failure of the right ventricle defined as the need for a RV Assist Device
* Septic condition
* Cerebral Disease
* Bleeding with a need for surgical intervention
* Pulmonary embolism
* Allergy to Heparin or any known coagulopathy
* Aortic regurgitation >II°
* Pregnancy
* Inclusion in another study or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-08; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Cardiac index | within 1 hour after device implantation

SECONDARY OUTCOMES:
Hemodynamic and metabolic parameters | until to hospital discharge
Mortality | within 30 and 180 days
device-related complications:hemolysis and major bleedings | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Melchior Seyfarth, MD, Study Chair — Deutsches Herzzentrum Muenchen; Josef Dirschinger, MD, Principal Investigator — 1. Medizinische Klinik, Klinikum rechts der Isar
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Hochman JS, Sleeper LA, Webb JG, Dzavik V, Buller CE, Aylward P, Col J, White HD; SHOCK Investigators. Early revascularization and long-term survival in cardiogenic shock complicating acute myocardial infarction. JAMA. 2006 Jun 7;295(21):2511-5. doi: 10.1001/jama.295.21.2511. PMID 16757723
- [Background] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Background] Ryan TJ, Antman EM, Brooks NH, Califf RM, Hillis LD, Hiratzka LF, Rapaport E, Riegel B, Russell RO, Smith EE 3rd, Weaver WD, Gibbons RJ, Alpert JS, Eagle KA, Gardner TJ, Garson A Jr, Gregoratos G, Ryan TJ, Smith SC Jr. 1999 update: ACC/AHA guidelines for the management of patients with acute myocardial infarction. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on Management of Acute Myocardial Infarction). J Am Coll Cardiol. 1999 Sep;34(3):890-911. doi: 10.1016/s0735-1097(99)00351-4. No abstract available. PMID 10483976
- [Derived] Seyfarth M, Sibbing D, Bauer I, Frohlich G, Bott-Flugel L, Byrne R, Dirschinger J, Kastrati A, Schomig A. A randomized clinical trial to evaluate the safety and efficacy of a percutaneous left ventricular assist device versus intra-aortic balloon pumping for treatment of cardiogenic shock caused by myocardial infarction. J Am Coll Cardiol. 2008 Nov 4;52(19):1584-8. doi: 10.1016/j.jacc.2008.05.065. PMID 19007597